CLINICAL TRIAL: NCT01864980
Title: Monitoring of Intraoperative Blood Loss: Benefit of Continuous Noninvasive Haemoglobin Monitoring?
Brief Title: Intra-operative Monitoring of Blood Loss
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof.dr.T.W.L.Scheeren, Prof.dr., University Medical Center Groningen
Other Study IDs: bleeding SpHb-001
Record Dates: First submitted 2013-05-22; First posted 2013-05-30 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Undetected Intraoperative Blood Loss
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hb group:15 patients: scheduled for elective surgery associated with undetected, i.e., difficult to reliably monitor intraoperative blood loss.
  Interventions: Procedure: blood transfusion, intermittent Hbsatlab measurement
- SpHb group: 15 patients: scheduled for elective surgery associated with undetected, i.e., difficult to reliably monitor intraoperative blood loss.
  Interventions: Procedure: blood transfusion, based on continuous SpHb readings

INTERVENTIONS:
Procedure: blood transfusion, intermittent Hbsatlab measurement — In the Hbsatlab group, RBC administration and its timing will be based on intermittent Hbsatlab measurement (routine care)
  Groups: Hb group:15 patients
Procedure: blood transfusion, based on continuous SpHb readings — RBC administration and its timing will be based on continuous SpHb readings while Hbsatlab values, measured every 30 min. by an objective observer, will not be visible to the attending anaesthetist.
  Groups: SpHb group: 15 patients

SUMMARY:
Certain types of surgery are associated with occult blood loss, which is hard to detect intraoperatively by intermittent conventional, invasive Hb concentration measurements using the clinical standard of Hb monitoring by satellite laboratory analysis (Hbsatlab). The investigators want to see whether continuous non-invasive transcutaneous Hb measurement using a finger sensor (SpHb), (a) reduces the total time (area under the curve, AUC) a patient's Hb is below a predetermined transfusion threshold (HbAUC) for administration of red blood cell concentrate (RBC), and (b) prevents a decrease in total oxygen delivery (DO2) possibly associated with transfusion below a critical haemoglobin concentration. Furthermore, the investigators want to study if SpHb monitoring changes the timing of RBC administration and reduces the need for intra- and post-operative RBC transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the age of 18 years or older, planned for elective surgery at-risk for undetected blood loss.
* American Society of Anesthesiologists (ASA) classification I, II, III, IV

Exclusion Criteria:

* Patient refusal
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 adult patients scheduled for surgery associated with undetected, i.e., difficult to reliably monitor intraoperative blood loss
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
HbAUC | during operation
  the total time a patient's Hb is below a predetermined transfusion threshold (HbAUC) for administration of red blood cell concentrate

SECONDARY OUTCOMES:
blood transfusions | intra- and post operative up to 48h
  the number of perioperative blood transfusions

OTHER OUTCOMES:
DO2 | intraoperative
  DO2 = oxygen delivery
serum concentrations of high-sensitive troponin T | post operative up to 48h
  serum concentrations of high-sensitive troponin T
serum concentrations of lactate | intra- and post operative up to 48h
  lactate
StO2 | intraoperative
  StO2 = peripheral tissue oxygenation by near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Michel M.R.F. Struys, Prof.dr, Principal Investigator — University of groningen,University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands